CLINICAL TRIAL: NCT03185195
Title: An Open-Label,2-Part Sequential Dose Study Designed to Assess the Absolute Bioavailability, Mass Balance Recovery, Metabolite Profile and Identification of Metabolite Structure for [14C]-AQX-1125 in Healthy Subjects
Brief Title: Phase 1 Absorption Distribution Metabolism and Excretion of AQX-1125
Acronym: ADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aquinox Pharmaceuticals (Canada) Inc. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AQX-1125-103
Record Dates: First submitted 2017-03-08; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 4-(4-(aminomethyl)-7a-methyl-1-methylideneoctahydro-1H-inden-5-yl)-3-(hydroxymethyl)-4-methylcyclohexan-1-ol

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- AQX-1125 Oral Tablet (Experimental): AQX-1125 - Oral Tablet
  Interventions: Drug: AQX-1125 Oral Tablet
- [14C]-AQX-1125 IV (Experimental): Radiolabelled AQX-1125 - Intravenous
  Interventions: Drug: [14C]-AQX-1125 IV
- [14C]-AQX-1125 Oral Solution (Experimental): Radiolabelled AQX-1125 - Oral Solution
  Interventions: Drug: [14C]-AQX-1125 Oral Solution

INTERVENTIONS:
Drug: AQX-1125 Oral Tablet — Part 1: Subjects will receive a single oral dose of AQX-1125 followed by [14C]-AQX-1125 IV Microtracer dose. In Part 2 subjects receive [14C]-AQX-1125 oral solution.
  Arms: AQX-1125 Oral Tablet
Drug: [14C]-AQX-1125 IV — Part 1: Subjects will receive a single oral dose of AQX-1125 followed by [14C]-AQX-1125 IV Microtracer dose. In Part 2 subjects receive [14C]-AQX-1125 oral solution.
  Other Names: Radiolabelled AQX-1125 IV
  Arms: [14C]-AQX-1125 IV
Drug: [14C]-AQX-1125 Oral Solution — Part 1: Subjects will receive a single oral dose of AQX-1125 followed by [14C]-AQX-1125 IV Microtracer dose. In Part 2 subjects receive [14C]-AQX-1125 oral solution.
  Other Names: Radiolabelled AQX-1125 Oral Solution
  Arms: [14C]-AQX-1125 Oral Solution

SUMMARY:
This study is conducted to evaluate the absolute bioavailability, metabolism and elimination pathways of AQX-1125 in healthy male and female subjects.

DETAILED DESCRIPTION:
This is a single-centre, open-label, non-randomised, 2-part, sequential dose study in healthy male and female subjects. It is planned to enrol a single cohort of 8 healthy subjects (4 male and 4 female) who will participate in Part 1 and Part 2 of the study.

In Part 1, each subject will receive a single oral dose of AQX-1125 followed by an IV microtracer dose of carbon-14-AQX-1125 ([14C]-AQX-1125). In Part 2, each subject will receive a single oral dose of [14C]-AQX-1125.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Healthy females of non-child bearing potential
* BMI 18.0 to 35 kg/m2

Exclusion Criteria:

* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who had smoked within the last 12 months; this included cigarettes, e-cigarettes and nicotine replacement products. Positive cotinine test result at screening and each admission
* Clinically significant abnormal clinical chemistry, haematology, urinalysis or electrocardiogram (ECG)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Absolute bioavailability (F) of AQX-1125 | 0 - 96 hrs
Mass balance recovery of total radioactivity in urine, faeces and all excreta | 0 -168 hrs
  Measure amount excreted (Ae)
Mass balance recovery of total radioactivity in urine, faeces and all excreta | 0 -168 hrs
  Measure Ae as a percentage of the administered dose (%Ae)
Mass balance recovery of total radioactivity in urine, faeces and all excreta | 0 -168 hrs
  Cumulative recovery of Ae (Cum Ae)
Mass balance recovery of total radioactivity in urine, faeces and all excreta | 0 -168 hrs
  Cum Ae expressed as a percentage of the administered dose (Cum %Ae)
Metabolite profiling and structural identification in plasma, urine and faeces to estimate the routes and rates of elimination of [14-C]-AQX-1125 | 0 -168 hrs
Measure Ae total radioactivity for urine and faeces | 0-168 hrs
Measure %Ae total radioactivity for urine and faeces | 0-168 hrs
Measure Cum Ae (total) for urine and faeces | 0-168 hrs
Measure Cum% Ae (total) for urine and faeces | 0-168 hrs
Measure PK parameters of total radioactivity in plasma following oral administration | 0 -96 hrs
  Cmax
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  Tmax
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  Tlag
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  AUC (0-24)
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  AUC (0-last)
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  AUC (0-inf)
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  AUC % extrap
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  lambda-z
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  T1/2
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  CL/F
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  Vz/F
Measure PK parameters of total radioactivity in plasma following oral administration: | 0 -96 hrs
  MRT

SECONDARY OUTCOMES:
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of Cmax
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of Tmax
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of Tlag
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of AUC(0-24)
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of AUC(0-last)
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of AUC(0-inf)
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of AUC%extrap
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of lambda-z
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of T1/2
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of CL/F
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of Vz/F
PK parameters of AQX-1125 in plasma following oral administration (Part 1) | 0-96 hrs
  Measurement of MRT
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of Cmax
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of Tmax
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of Tlag
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of AUC(0-24)
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of AUC(0-last)
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of AUC(0-inf)
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of AUC%extrap
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of lambda-z
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of T1/2
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of CL
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of Vz
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of VSS
PK parameters of AQX-1125 in plasma following IV administration (Part 1) | 0 - 96 hrs
  Measurement of MRT
Safety and tolerability assessments based on adverse events, safety laboratory tests, vital signs, physical examinations, ECGs and AEs (Part 1) | 0 - 96 hrs
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of Cmax
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of Tmax
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of Tlag
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of AUC(0-24)
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of AUC(0-last)
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of AUC(0-inf)
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of AUC%extrap
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of lambda-z
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of T1/2
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of CL/F
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of Vz/F
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of F
PK parameters of AQX-1125 in plasma following oral administration (Part 2) | 0 -168 hrs
  Measurement of MRT
Measure plasma whole blood concentration ratios for total radioactivity (Part 2) | 0 -168 hrs
Chemical structure of major metabolites of [14-C]-AQX-1125 | 0 -168 hrs
  Major metabolites classified as >10% of the AUC of total radioactivity in plasma and >10% dose excreted in urine and faeces following oral administration (Part 2)
Safety and tolerability assessments based on adverse events, safety laboratory tests, vital signs and ECG (Part 2) | 0 -168 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Nand Singh, MD, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No